CLINICAL TRIAL: NCT03008590
Title: Low Dose Naltrexone for Chronic Pain in Osteoarthritis and Inflammatory Arthritis
Brief Title: Low Dose Naltrexone for Chronic Pain From Arthritis
Acronym: LDN-VA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NURB-008-16S
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic
Keywords: Pain management; Naltrexone; Controlled clinical trials, randomized
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic; Agnosia | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone first then placebo (Other): Naltrexone for 8 weeks, then placebo for 8 weeks, blinded cross-over design
  Interventions: Drug: Naltrexone; Drug: Placebo
- Placebo first then naltrexone (Other): Placebo for 8 weeks, then naltrexone for 8 weeks, blinded cross-over design
  Interventions: Drug: Naltrexone; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — One 4.5 mg capsule each evening
Drug: Placebo — One capsule each evening

SUMMARY:
Over 100 million Americans report chronic pain. Veterans are disproportionately affected for multiple reasons, including injuries and post-traumatic stress disorder. Treatment for chronic pain is a priority research area for the VA. One of the most common causes of chronic pain is osteoarthritis (OA). OA is attributable to "wear and tear," but reasons for pain are complex. Inflammatory arthritis (IA) includes multiple severe diseases that affect 2-3% of persons and require treatment with immune-suppressive drugs to prevent joint destruction. Pain often persists despite effective treatment. Pain in arthritis results from multiple sources: inflammation, perception of pain in the joint, and interpretation of pain by the brain. Unfortunately, management of pain in arthritis remains a challenge. Low dose naltrexone is a widely used but unproven "alternative" approach to chronic pain. It is attractive for study because it is safe and is proposed to work on all three pathways that contribute to pain. A small but high-quality clinical trial is needed to determine whether to invest in definitive studies.

DETAILED DESCRIPTION:
Chronic pain affects over 100 million Americans, and arthritis is the most common cause. Existing treatments for chronic arthritic pain are only mildly effective, and risks of medications used to treat pain are numerous and continue to be discovered. Treatment of chronic is a high priority research area for VA CSR&D.

Naltrexone is an opioid antagonist that is FDA approved in an oral daily dose of 50 mg to prevent recidivism in alcoholics. At much lower doses of 4 - 4.5 mg daily, however, it has been shown in small, blinded, randomized trials to improve pain in fibromyalgia, gastrointestinal symptoms in Crohn's disease, and quality of life in multiple sclerosis. The only other published data are case reports in complex regional pain syndrome, low back pain, and scleroderma. However, advocacy of low-dose naltrexone (LDN) by internet-based MDs and patients is high, and since LDN can be prescribed off-label, its use greatly exceeds what is justified by evidence. The drug can be prescribed only via compounding pharmacies, so its use costs a patient ~$40/month.

Among the many unproven treatments that are widely used, LDN is of particular interest because results of surveys of patients are particularly impressive, because it is quite safe, and because its benefit is plausible pharmacologically. There is evidence both for modulation of central pain-processing pathways and for down-regulation of inflammatory pathways in microglia. Considering the diversity of conditions proposed to benefit from LDN and the unequivocal need for better approaches to pain relief in chronic conditions, high-quality clinical trials are needed in both inflammatory and non-inflammatory conditions. This small but placebo-controlled study, powered to detect an effect size as small as that seen with NSAIDs or the most beneficial non-pharmacologic approaches, is proposed as a prerequisite for considering a pivotal trial through the VA Cooperative Studies Program.

The proposed study is a randomized, double-blinded, cross-over, placebo-controlled trial in adults with osteoarthritis or inflammatory arthritis and persistent pain. Sixty patients will be enrolled for 16 weeks, during which they will receive LDN for 8 weeks and placebo for 8 weeks. Widely accepted patient-reported outcome measures will be used. The co-primary endpoints are reduction in pain severity or pain's interference with function during 8 weeks of LDN compared to 8 weeks placebo, using the Brief Pain Inventory. Other patient-reported data will be used both as secondary outcomes and as covariates in analyzing determinants of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria in order to be eligible for enrollment:

* Veteran or otherwise eligible for VA benefits, able to travel to VA Boston
* One or more of the following chronic conditions:

  * osteoarthritis
  * rheumatoid arthritis
  * non-axial spondyloarthritis
* Average daily pain interference with function (average of the 7 parts of question 9 on the Brief Pain Inventory) rated at least 4 on a scale of 0-10, and no higher than 9
* No change in medication in the past 8 weeks made with the expectation of improving pain
* No plan to start another medication or a non-pharmacologic treatment regimen likely to affect pain during the next 16 weeks
* Age at least 18
* Registered for medical care in the VA Boston Healthcare System
* Capable of informed consent, and willingness to comply with study procedures, including receipt of weekly phone calls from the study coordinator

Exclusion Criteria:

Any of the following requires exclusion from participation:

* Current use of opioids including tramadol
* Pregnant, breast feeding, or unwilling to engage in contraceptive practices if sexually active and capable of conceiving
* Schizophrenia, bipolar disorder, or poorly controlled depression or anxiety
* Previous use of low-dose naltrexone
* Back pain described by the patient as greater in severity than arthritic pain in a non-axial location
* Significant kidney disease, defined as glomerular filtration rate < 30 ml/min
* Liver cirrhosis. There is no specific screening procedure to exclude cirrhosis.
* Painful peripheral neuropathy. There is no specific screening procedure.
* Plan to have surgery during the next 16 weeks
* Inconsistency in self-reporting at the screening visit. BPI, PainDETECT, WOMAC, and PROMIS-29 all contain 0-10 scales of average pain intensity, although the times listed vary from 1-4 weeks. The severity reported on these three scales cannot differ by more than 1.
* Other qualitative circumstances that the investigator feels would make the patient a poor candidate for this clinical trial, such as an unstable social situation or unreliable transportation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Monach, MD PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset containing all the primary study data will be created and shared per VA policies. This dataset will be included as a supplementary file attached to the published manuscript, which in turn will be available through PubMed Central per VA rules. In the event that the study has not been published, the dataset will be made available by other means within 3 years of study completion. The publicly available dataset will not include any identifiers, e.g. age will be included but not birthdate.
Supporting Information: ICF
Time Frame: ICF to be posted within 3 months per VA policy. De-identified dataset to be included as supplementary material with publication, anticipated to be within 12 months of study completion.

REFERENCES:
- [Derived] Beaudette-Zlatanova B, Lew RA, Otis JD, Branch-Elliman W, Bacorro E, Dubreuil M, Eyvazzadeh C, Kaur M, Lazzari AA, Libbey C, Monach PA. Pilot Study of Low-dose Naltrexone for the Treatment of Chronic Pain Due to Arthritis: A Randomized, Double-blind, Placebo-controlled, Crossover Clinical Trial. Clin Ther. 2023 May;45(5):468-477. doi: 10.1016/j.clinthera.2023.03.013. Epub 2023 Apr 10. PMID 37045708

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone First Then Placebo | Placebo First Then Naltrexone
Started | 14 | 15
Completed | 11 | 12
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Patients who completed the study
Groups:
- Naltrexone First: Received naltrexone first, then placebo
- Placebo First: Received placebo first, then naltrexone
- Total: Total of all reporting groups
Arm/Group | Naltrexone First | Placebo First | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.2) | 64 (11.9) | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23
Diagnosis, OA or IA [Count of Participants; unit: Participants]
  Osteoarthritis | 7 | 10 | 17
  Inflammatory arthritis | 4 | 2 | 6
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33 (7.9) | 35 (6.9) | 34 (7.3)
Brief Pain Inventory - Pain interference (sum of 7 subscales, each 0-10) [Mean (Standard Deviation); unit: units on a 0-70 scale (higher is worse)] | 39 (9.5) | 42 (11.5) | 41 (10.5)
Brief Pain Inventory - Pain severity [Mean (Standard Deviation); unit: units on a 0-10 scale (higher is worse)] | 5.9 (1.2) | 5.9 (1.3) | 5.9 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory - Pain Interference
Description: Sum of 7 questions (each on a 0-10 scale, therefore 0-70 total) on how much pain has interfered with general function, walking ability, mood, normal work, relations with other people, sleep, and enjoyment of life. Higher score is a worse outcome. Results are reported as change from baseline: after 8 weeks of naltrexone, or after 8 weeks of placebo.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone or 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- At End of 8 Weeks Naltrexone Treatment; At End of 8 Weeks Placebo Treatment: Data from naltrexone periods were pooled for presentation purposes, but period (first or second) was included as a variable in the statistical analysis. Results shown are change from baseline.
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -23 (19.4) | -22 (19.2)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; Data from the primary or secondary outcome measures were the dependent variables. The patient was the random effect. Dependent fixed effects variables included treatment at the time of data collection (naltrexone or placebo), group (naltrexone first or placebo first), and week (4, 8, 12, and 16); Test type: Superiority; p = 0.90, Mixed Models Analysis — Significance pre-specified at P<0.05

2. Secondary Outcome: Brief Pain Inventory - Pain Severity
Description: Average severity of pain in the past 7 days (0-10). Higher score is a worse outcome. Results are reported as change from baseline: after 8 weeks naltrexone, and after 8 weeks placebo.
Time Frame: 8 and16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -1.7 (1.87) | -2.0 (2.17)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.22, Mixed Models Analysis — Significance pre-specified at P<0.05

3. Secondary Outcome: painDETECT
Description: Measure of neuropathic pain (0-38). Lower score indicates nociceptive pain, higher score indicates neuropathic pain. Results are reported as change from baseline: after 8 weeks of naltrexone or after 8 weeks placebo.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -4.0 (6.26) | -5.6 (5.73)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02, Mixed Models Analysis — Although significance was pre-specified at P<0.05, it is suspected that this result is spurious due to multiple comparisons

4. Secondary Outcome: Brief Fatigue Inventory
Description: Questionnaire, severity of fatigue and fatigue's interference with activity (0-10 scales). Higher score is a worse outcome. Results are reported as change from baseline: after 8 weeks naltrexone or after 8 weeks placebo.
Time Frame: 8 and16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -1.8 (1.61) | -1.8 (2.71)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3, Mixed Models Analysis — Significance pre-specified at P<0.05

5. Secondary Outcome: Beck Depression Inventory-II
Description: Questionnaire measuring severity of depression (0-69). Used primarily during screening to exclude enrollment of patients with severe depression, but also as a safety outcome measure during the study. Higher score is a worse outcome. Results are reported as change from baseline: after 8 weeks of naltrexone, or after 8 weeks of placebo
Time Frame: 8 and16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -1.0 (4.29) | -1.7 (6.04)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Clinical Global Impression of Severity (CGI-S)
Description: 7-point scale (1-7) of patients' self-reporting of severity during the study. Higher score is a worse outcome. Results are reported as change from baseline: after 8 weeks naltrexone, or after 8 weeks placebo.
Time Frame: 8 and16 weeks, ie after 8 weeks naltrexone and 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -1.1 (1.59) | -1.1 (1.83)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.78, Mixed Models Analysis — Significance pre-specified at P<0.05

7. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I)
Description: 7-point scale (1-7) of patients' self-reporting of improvement or worsening during the study. A higher score is a worse outcome. Results are reported as change from baseline: after 8 weeks naltrexone, or after 8 weeks placebo.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 23 | 23
units on a scale | -0.3 (1.2) | -0.2 (1.71)
Statistical Analysis 1: Comparison: At End of 8 Weeks Naltrexone Treatment vs At End of 8 Weeks Placebo Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.92, Mixed Models Analysis — Significance pre-specified at P<0.05

8. Secondary Outcome: Patient Reported Outcomes Measurement Information System Profile (PROMIS-29)
Description: Questionnaire, survey of 29 questions assessing health-related quality of life across 8 domains. The subscores are not added to give a single score. Results would have been reported as change from baseline (after 8 weeks naltrexone, or after 8 weeks placebo), but data were not collected.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Population: Data not collected
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: C Reactive Protein (CRP)
Description: Blood test for inflammation. Plan was to reported as change from baseline (after 8 weeks naltrexone, or after 8 weeks placebo), but data were not collected.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Population: Data were not collected
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Disease Activity Score (DAS28)
Description: Measure of disease activity in rheumatoid arthritis. Plan was to reported report results as change from baseline (after 8 weeks naltrexone, or after 8 weeks placebo), but data were not collected.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Population: Data not collected.
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Bath Ankylosing Spondylitis Activity Index (BASDAI)
Description: Patient-reported index of disease activity for ankylosing spondylitis. Higher is more severe. Results would have been reported as change from baseline (after 8 weeks naltrexone, or after 8 weeks placebo) but data were not collected.
Time Frame: 8 and 16 weeks, ie after 8 weeks naltrexone and after 8 weeks placebo
Population: Data not collected
Arm/Group | At End of 8 Weeks Naltrexone Treatment | At End of 8 Weeks Placebo Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks (8 weeks each naltrexone and placebo)
Groups:
- During Naltrexone Treatment: Adverse events during naltrexone
- During Placebo Treatment: Adverse events during placebo
Arm/Group | During Naltrexone Treatment | During Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/29
Other Adverse Events (participants affected / at risk) | 7/29 | 12/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | During Naltrexone Treatment (N=29) | During Placebo Treatment (N=29)
Anaplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Shortness of breath of unknown origin, led to hospitalization, resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | During Naltrexone Treatment (N=29) | During Placebo Treatment (N=29)
Fatigue (General disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Infections, minor viral or bacterial (Infections and infestations) | 1 (1) | 5 (5)
Abdominal / GI symptoms (Gastrointestinal disorders) | 0 (0) | 3 (3) — Nausea, vomiting, bloating
Lip and tongue swelling (Immune system disorders) | 1 (1) | 0 (0) — Suspected allergic reaction
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — One case poison ivy, another unknown, both resolved
Reduced renal function (Renal and urinary disorders) | 0 (0) | 1 (1) — Mild, transient reduction in GFR, unknown cause
Ankle injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT03008590/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03008590/Prot_SAP_001.pdf